CLINICAL TRIAL: NCT00874991
Title: Cardiac Deformation: Correlation With Conventional Echocardiographic Hemodynamic Variables. An Intraoperative Study.
Brief Title: Cardiac Deformation: Correlation With Conventional Echocardiographic Hemodynamic Variables (An Intraoperative Study)
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 0709009426
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Cardiac Disease
Keywords: Cardiac deformation; Cardiopulmonary bypass; TEE; Cardiac Surgery; Left ventricular function; Pulmonary Artery catheter; Tissue Doppler; Left ventricular function in cardiac surgery
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this research is to apply cardiac tissue characterization in order to assess left ventricular function in cardiac surgical patients pre and post cardiopulmonary bypass. The procedures to be used include a retrospective review of transesophageal images obtained during conventional intraoperative transesophageal echocardiography (TEE) for cardiac surgery, as well as a secondary analysis with Tissue Doppler. The results will be compared with hemodynamic data obtained from a pulmonary artery catheter (PAC).

DETAILED DESCRIPTION:
Patients included in this study are between the ages of 18 to 99 years of age, who presented to the operating room for cardiac surgery, and received both a pulmonary artery catheter and a routine intra-operative TEE. We will only be looking at patients whose TEE images were of good quality.

Subjects underwent cardiac surgery and received both a PAC and a routine TEE exam. We will review the data from the PAC, the images from the conventional TEE exam, and a secondary analysis with Tissue Doppler.

A potential benefit to society is a novel means for assessing left ventricular function. Our research will not benefit our subjects directly. There is no additional risk to our subjects beyond the insertion of the PAC and the TEE probe, which are routinely placed in our patients under-going cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients >18 years of age Patients scheduled for cardiac surgery and will receive both a pulmonary artery catheter and a routine intra-operative TEE

Exclusion Criteria:

* TEE images that are of poor quality

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery with general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2008-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
assess left ventricular function in cardiac patients pre and post cardiopulmonary bypass | 1

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Skubas, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD